CLINICAL TRIAL: NCT04375254
Title: The Effect of the Use Of Neuroscience-based Nomenclature (NbN) In The Teaching Of Psychopharmacology on Medical Students Views Toward Psychiatry
Brief Title: Neuroscience-based Nomenclature (NbN) as a Teaching Tool
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Jerusalem Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Daniel Minkin Levy, Psychiatry clerkship clinical guide, Hebrew University of Jerusalem
Other Study IDs: 0103wrqw2030
Record Dates: First submitted 2020-05-03; First posted 2020-05-05 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Medical Education
Keywords: psychopharmacology; students views on psychiatry; medical education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Medical students during psychiatry clerkship who received NbN psychopharmacology training
  Interventions: Other: NbB psychopharmacology training
- Control group: Medical students during psychiatry clerkship who received standard psychopharmacology training

INTERVENTIONS:
Other: NbB psychopharmacology training — a two part course in psychopharmacology based on Neuroscience based Nomenclature
  Groups: Intervention group

SUMMARY:
In recent decades, medical student interest in a career in mental health appear to be in decline, possibly due to the perception that the scientific foundation of psychiatry and psychopharmacology is weaker compared to other fields of medicine.

In an effort to examine ways of improving the current nomenclature in Psychopharmacology, in 2008 the nomenclature taskforce was initiated, composed of representatives from five international organizations: ECNP - European College of Neuropsychopharmacology, ACNP - American College of Neuropsychopharmacology, AsCNP - Asian College of Neuropsychopharmacology, CINP - International College of Neuropsychopharmacology, IUPHAR - International Union of Basic and Clinical Pharmacology.2 The result of this effort is the Neuroscience based Nomenclature (NbN) - a pharmacologically driven nomenclature that focuses on reflecting current knowledge and on the understanding of the neural system being modified

this research is the first that examine whether putting greater emphasis on neuroscience in the teaching of psychotropics, through the use of the new NbN terminology, achieve the goal of improving medical students views on psychiatry.

DETAILED DESCRIPTION:
In recent decades, medical student interest in a career in mental health appear to be in decline1. There are multiple factors responsible for the apparent lack of interest in psychiatry, one of them may be the perception that the scientific foundation of psychiatry and psychopharmacology is weaker compared to other fields of medicine.

As the field of psychopharmacology evolves, the terminology used to describe different classes of medication becomes increasingly convoluted: at a time when the same agent is used for the treatment of several different disorders, the nomenclature in use is indication-based and divided into classes that are disease based - such as Antidepressant, Antipsychotic and Anxiolytics. These classes, in turn, are divided into subclasses like "Atypical" or "Second Generation" - terms that give little information regarding the pharmacological properties of the medication itself.

This discrepancy between the current naming of psychotropics and the way they are used in clinical practice is confusing to both the clinician and the patient - and since it fails to reflect on the current scientific knowledge, may affect the way young medical professionals perceive the profession of psychiatry.

In an effort to examine ways of improving the current nomenclature in Psychopharmacology, in 2008 the nomenclature taskforce was initiated, composed of representatives from five international organizations: ECNP - European College of Neuropsychopharmacology, ACNP - American College of Neuropsychopharmacology, AsCNP - Asian College of Neuropsychopharmacology, CINP - International College of Neuropsychopharmacology, IUPHAR - International Union of Basic and Clinical Pharmacology.2 The result of this effort is the Neuroscience based Nomenclature (NbN) - a pharmacologically driven nomenclature that focuses on reflecting current knowledge and on the understanding of the neural system being modified (''pharmacological domain'') and its mode/mechanism of action (''mode of action'')3. The NbN was widely accepted by both clinicians and leading psychiatric journals4 The need to revise the teaching methods of psychopharmacology was reviewed over the years, with different strategies suggested5. To our knowledge, this research is the first that examine whether putting greater emphasis on neuroscience in the teaching of psychotropics, through the use of a new terminology, achieve the goal of improving medical students views on psychiatry.

ELIGIBILITY:
Inclusion Criteria:

Medical students during fifth year psychiatry clerkship

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical students during fifth year psychiatry clerkship
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
NbN influence on medical students views on psychiatry | May-September 2020
  To examine if Neuroscience-based Nomenclature (NbN) as a teaching-tool for medical students affects their views about the scientific foundation of psychiatry and psychopharmacology.

SECONDARY OUTCOMES:
NbN influence on choosing psychiatry as a profession | May-September 2020
  To examine whether the use of Neuroscience-based Nomenclature (NbN) in the teaching of psychopharmacology can improve medical students' views on choosing a career in psychiatry.

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Joseph, MD, Study Director — Haim Sheba Medical Center
Locations (1):
- Jerusalem Center for Mental Health, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tamaskar P, McGinnis RA. Declining student interest in psychiatry. JAMA. 2002 Apr 10;287(14):1859. No abstract available. PMID 11939877
- [Background] Zohar J, Nutt DJ, Kupfer DJ, Moller HJ, Yamawaki S, Spedding M, Stahl SM. A proposal for an updated neuropsychopharmacological nomenclature. Eur Neuropsychopharmacol. 2014 Jul;24(7):1005-14. doi: 10.1016/j.euroneuro.2013.08.004. Epub 2013 Sep 18. PMID 24630385
- [Background] Zohar J, Kasper S. Neuroscience-based Nomenclature (NbN): A call for action. World J Biol Psychiatry. 2016 Aug;17(5):318-20. doi: 10.1080/15622975.2016.1193626. Epub 2016 Jul 5. No abstract available. PMID 27379490
- [Background] The Lancet Psychiatry. Naming names. Lancet Psychiatry. 2016 Jun;3(6):489. doi: 10.1016/S2215-0366(16)30072-4. No abstract available. PMID 27262036
- [Background] Zisook S, Glick ID, Jefferson JW, Wagner KD, Salzman C, Peselow ED, Stahl S. Teaching psychopharmacology: what works and what doesn't. J Clin Psychopharmacol. 2008 Feb;28(1):96-100. doi: 10.1097/jcp.0b013e3181603f6b. PMID 18204350